CLINICAL TRIAL: NCT01491919
Title: Safety and Pharmacokinetics of Lisinopril in Pediatric Kidney Transplant Recipients
Brief Title: Safety Study of Lisinopril in Children and Adolescents With a Kidney Transplant
Acronym: PTN_LISINO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Uptal Patel (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); The Emmes Company, LLC (Industry); University of Rochester (Other); OpAns, LLC (Unknown)
Responsible Party: Sponsor-Investigator, Uptal Patel, Assoc Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00029537; HHSN275201000003I (Other: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD))
Record Dates: First submitted 2011-11-29; First posted 2011-12-14 (Estimated); Results first posted 2015-07-08 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-06

CONDITIONS: Hypertension
Keywords: High Blood Pressure; Hypertension; Renal Transplantation; Kidney Transplantation
MeSH Terms: conditions — Hypertension | interventions — Lisinopril

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low Dose: Lisinopril (Experimental): Participants will receive study medication for 14±3 days at a dose 0.1 mg/kg/day
  Interventions: Drug: Lisinopril
- Medium Dose: Lisinopril (Experimental): Participants will receive study medication for 14±3 days at a dose 0.2 mg/kg/day
  Interventions: Drug: Lisinopril
- High Dose: Lisinopril (Experimental): Participants will initially receive study medication at 0.2 mg/kg/day for 5±2 days. If blood tests exclude drug-related toxicity, then the lisinopril dose will be increased to 0.4 mg/kg/day and participants will continue to complete the 14±3 day Treatment Period.
  Interventions: Drug: Lisinopril

INTERVENTIONS:
Drug: Lisinopril — Subjects will be randomized to Low, Medium, or High dose of Lisinopril

SUMMARY:
The drug lisinopril is approved by the U.S. Food and Drug Administration for the treatment of high blood pressure, heart failure, and acute heart attacks in adult patients. In children over 6 years of age, lisinopril is approved for the treatment of high blood pressure. Lisinopril is in a group of medications called angiotensin-converting enzyme inhibitors (ACE). ACE inhibitors such as lisinopril work by decreasing certain chemicals that tighten the blood vessels so blood flows more smoothly and the heart can pump blood more efficiently.

There is some information available about how children with high blood pressure absorb, distribute, metabolize, and eliminate lisinopril (this information about medication processing by the body is called pharmacokinetic data). However, there is no information about how children with high blood pressure who have received a kidney transplant process lisinopril. In addition to decreasing blood pressure, investigators believe that lisinopril may help kidney transplants work longer by reducing the activity of chemicals made by cells in kidney transplants that can lead to inflammation and injury. Such benefits have not been found with another group of blood pressure medications called calcium channel blockers, which are the most commonly used medication group to control high blood pressure in children after a kidney transplant. A clinical trial will be conducted in the future to compare which medication group helps kidney transplants in children last longer. To guide the selection of the best dose to test in future studies, investigators in this study will try to determine the safety profile, dose tolerability, and pharmacokinetics of lisinopril in children and adolescents (2-17 years of age) who have received a kidney transplant and have high blood pressure.

ELIGIBILITY:
Inclusion Criteria:

1. Kidney transplant recipient
2. Age 2-17 years, inclusive, at the time of first study dose
3. Estimated GFR (eGFR) ≥30 ml/min/1.73m2, with stable allograft function as indicated by <20% change in serum creatinine in the previous 30 days
4. Stable immunosuppressive regimen, as indicated by <10% change in dosage (in mg/kg) in these medications, within the 14 days prior to enrollment
5. Systolic BP >90th percentile for age, gender, and height, necessitating initiation or addition of an antihypertensive medication
6. For females of child-bearing potential, a negative serum pregnancy test prior to initial dosing and agreement to practice appropriate contraceptive measures, including abstinence, from the time of the initial pregnancy testing through the remainder of the study (30 days after last administration of investigational agents).

Exclusion Criteria:

1. History of anaphylaxis attributable to lisinopril or other angiotensin-converting enzyme inhibitor (ACEI) agents (e.g.,enalapril, ramipril, quinapril)
2. History of anaphylaxis attributable to iohexol or an iodine hypersensitivity
3. Use of an angiotensin-converting enzyme inhibitor (ACEI), angiotensin receptor blocker, or renin antagonist within 30 days prior to enrollment
4. Stage 2 hypertension defined as the >99th percentile for age, height and gender + 5 mm Hg
5. Blood Potassium value > 6.0 milliequivalent / liter (mEq/L) (as determined at the screening visit)
6. Previous participation in this study
7. Physician concern that the participant may not adhere to the study protocol, based on prior behavior
8. Current plasmapheresis treatment
9. History of angioedema
10. Pregnancy

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2012-06; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Benjamin, MD, PhD, MPH, Study Director — Duke University; Howard Trachtman, MD, Study Chair — NYU Langone Health; Uptal D Patel, MD, Principal Investigator — Duke University; Adam Frymoyer, MD, Principal Investigator — Stanford University
Locations (7):
- United States (7):
  - University of Alabama, Birmingham, Alabama
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Emory University and Children's Healthcare of Atlanta, Atlanta, Georgia
  - University of Michigan, Ann Arbor, Michigan
  - Children's Mercy Hospitals & Clinics, Kansas City, Missouri
  - New York University Langone Medical Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

REFERENCES:
- [Background] National High Blood Pressure Education Program Working Group on High Blood Pressure in Children and Adolescents. The fourth report on the diagnosis, evaluation, and treatment of high blood pressure in children and adolescents. Pediatrics. 2004 Aug;114(2 Suppl 4th Report):555-76. No abstract available. PMID 15286277
- [Background] Knutter I, Wollesky C, Kottra G, Hahn MG, Fischer W, Zebisch K, Neubert RH, Daniel H, Brandsch M. Transport of angiotensin-converting enzyme inhibitors by H+/peptide transporters revisited. J Pharmacol Exp Ther. 2008 Nov;327(2):432-41. doi: 10.1124/jpet.108.143339. Epub 2008 Aug 19. PMID 18713951
- [Background] Lin JH, Chen IW, Ulm EH, Duggan DE. Differential renal handling of angiotensin-converting enzyme inhibitors enalaprilat and lisinopril in rats. Drug Metab Dispos. 1988 May-Jun;16(3):392-6. PMID 2900730
- [Background] Hogg RJ, Delucchi A, Sakihara G, Wells TG, Tenney F, Batisky DL, Blumer JL, Vogt BA, Lo MW, Hand E, Panebianco D, Rippley R, Shaw W, Shahinfar S. A multicenter study of the pharmacokinetics of lisinopril in pediatric patients with hypertension. Pediatr Nephrol. 2007 May;22(5):695-701. doi: 10.1007/s00467-006-0399-5. Epub 2007 Jan 10. PMID 17216247
- [Background] Prinivil® (lisinopril tablets) package insert; Whitehouse Station, NJ: Merck & Co., Inc.; 2003
- [Background] Mitsnefes MM, Khoury PR, McEnery PT. Early posttransplantation hypertension and poor long-term renal allograft survival in pediatric patients. J Pediatr. 2003 Jul;143(1):98-103. doi: 10.1016/S0022-3476(03)00209-9. PMID 12915832
- [Background] Silverstein DM, Leblanc P, Hempe JM, Ramcharan T, Boudreaux JP. Tracking of blood pressure and its impact on graft function in pediatric renal transplant patients. Pediatr Transplant. 2007 Dec;11(8):860-7. doi: 10.1111/j.1399-3046.2007.00753.x. PMID 17976120
- [Background] Mitsnefes MM, Omoloja A, McEnery PT. Short-term pediatric renal transplant survival: blood pressure and allograft function. Pediatr Transplant. 2001 Jun;5(3):160-5. doi: 10.1034/j.1399-3046.2001.t01-1-00051.x. PMID 11422817
- [Background] Cross NB, Webster AC, Masson P, O'connell PJ, Craig JC. Antihypertensives for kidney transplant recipients: systematic review and meta-analysis of randomized controlled trials. Transplantation. 2009 Jul 15;88(1):7-18. doi: 10.1097/TP.0b013e3181a9e960. PMID 19584673
- [Background] Sorof JM, Goldstein SL, Brewer ED, Steiger HM, Portman RJ. Use of anti-hypertensive medications and post-transplant renal allograft function in children. Pediatr Transplant. 2000 Feb;4(1):21-7. doi: 10.1034/j.1399-3046.2000.00082.x. PMID 10731054
- [Background] Hernandez AA, Moreso F, Bayes B, Lauzurica R, Sanz-Guajardo D, Gomez-Huertas E, Pereira P, Paul J, Crespo J, Amenabar JJ, Oliver J, Seron D. Angiotensin-converting enzyme inhibitors and angiotensin receptor blockers in renal transplantation between 1990 and 2002 in Spain. NDT Plus. 2010 Jun;3(Suppl_2):ii21-ii25. doi: 10.1093/ndtplus/sfq068. PMID 20508862
- [Background] Mitterbauer C, Heinze G, Kainz A, Kramar R, Horl WH, Oberbauer R. ACE-inhibitor or AT2-antagonist therapy of renal transplant recipients is associated with an increase in serum potassium concentrations. Nephrol Dial Transplant. 2008 May;23(5):1742-6. doi: 10.1093/ndt/gfm864. Epub 2008 Jan 30. PMID 18234845
- [Background] Hiremath S, Fergusson D, Doucette S, Mulay AV, Knoll GA. Renin angiotensin system blockade in kidney transplantation: a systematic review of the evidence. Am J Transplant. 2007 Oct;7(10):2350-60. doi: 10.1111/j.1600-6143.2007.01928.x. PMID 17845569
- [Background] Morath C, Schmied B, Mehrabi A, Weitz J, Schmidt J, Werner J, Buchler MW, Morcos M, Nawroth PP, Schwenger V, Doehler B, Opelz G, Zeier M. Angiotensin-converting enzyme inhibitors and angiotensin II type 1 receptor blockers after renal transplantation. Clin Transplant. 2009 Dec;23 Suppl 21:33-6. doi: 10.1111/j.1399-0012.2009.01107.x. PMID 19930314
- [Background] Inigo P, Campistol JM, Lario S, Piera C, Campos B, Bescos M, Oppenheimer F, Rivera F. Effects of losartan and amlodipine on intrarenal hemodynamics and TGF-beta(1) plasma levels in a crossover trial in renal transplant recipients. J Am Soc Nephrol. 2001 Apr;12(4):822-827. doi: 10.1681/ASN.V124822. PMID 11274244
- [Background] Nielsen SE, Schjoedt KJ, Astrup AS, Tarnow L, Lajer M, Hansen PR, Parving HH, Rossing P. Neutrophil Gelatinase-Associated Lipocalin (NGAL) and Kidney Injury Molecule 1 (KIM1) in patients with diabetic nephropathy: a cross-sectional study and the effects of lisinopril. Diabet Med. 2010 Oct;27(10):1144-50. doi: 10.1111/j.1464-5491.2010.03083.x. PMID 20854382
- [Background] Halimi JM, Giraudeau B, Buchler M, Al-Najjar A, Etienne I, Laouad I, Bruyere F, Lebranchu Y. Enalapril/amlodipine combination in cyclosporine-treated renal transplant recipients: a prospective randomized trial. Clin Transplant. 2007 Mar-Apr;21(2):277-84. doi: 10.1111/j.1399-0012.2007.00643.x. PMID 17425758
- [Background] Spooner N, Lad R, Barfield M. Dried blood spots as a sample collection technique for the determination of pharmacokinetics in clinical studies: considerations for the validation of a quantitative bioanalytical method. Anal Chem. 2009 Feb 15;81(4):1557-63. doi: 10.1021/ac8022839. PMID 19154107
- [Background] Schwartz GJ, Munoz A, Schneider MF, Mak RH, Kaskel F, Warady BA, Furth SL. New equations to estimate GFR in children with CKD. J Am Soc Nephrol. 2009 Mar;20(3):629-37. doi: 10.1681/ASN.2008030287. Epub 2009 Jan 21. PMID 19158356
- [Background] Soffer B, Zhang Z, Miller K, Vogt BA, Shahinfar S. A double-blind, placebo-controlled, dose-response study of the effectiveness and safety of lisinopril for children with hypertension. Am J Hypertens. 2003 Oct;16(10):795-800. doi: 10.1016/s0895-7061(03)00900-2. PMID 14553956
- [Background] Thompson KC, Zhao Z, Mazakas JM, Beasley CA, Reed RA, Moser CL. Characterization of an extemporaneous liquid formulation of lisinopril. Am J Health Syst Pharm. 2003 Jan 1;60(1):69-74. doi: 10.1093/ajhp/60.1.69. PMID 12533979
- [Background] CDER Approval Package for Prinivil®: Application Number 19-558/S-043. Clinical Pharmacology and Biopharmaceutics Review. Available at: http://www.accessdata.fda.gov/drugsatfda_docs/nda/2003/19-558S043_Prinivil.cfm. Last accessed Jan. 6, 2011.
- [Background] Rhodin MM, Anderson BJ, Peters AM, Coulthard MG, Wilkins B, Cole M, Chatelut E, Grubb A, Veal GJ, Keir MJ, Holford NH. Human renal function maturation: a quantitative description using weight and postmenstrual age. Pediatr Nephrol. 2009 Jan;24(1):67-76. doi: 10.1007/s00467-008-0997-5. Epub 2008 Oct 10. PMID 18846389
- [Background] Thomson AH, Kelly JG, Whiting B. Lisinopril population pharmacokinetics in elderly and renal disease patients with hypertension. Br J Clin Pharmacol. 1989 Jan;27(1):57-65. doi: 10.1111/j.1365-2125.1989.tb05335.x. PMID 2539850
- [Background] Kuczmarski RJ, Ogden CL, Guo SS, Grummer-Strawn LM, Flegal KM, Mei Z, Wei R, Curtin LR, Roche AF, Johnson CL. 2000 CDC Growth Charts for the United States: methods and development. Vital Health Stat 11. 2002 May;(246):1-190. PMID 12043359
- [Background] Bazzoli C, Retout S, Mentre F. Design evaluation and optimisation in multiple response nonlinear mixed effect models: PFIM 3.0. Comput Methods Programs Biomed. 2010 Apr;98(1):55-65. doi: 10.1016/j.cmpb.2009.09.012. Epub 2009 Nov 4. PMID 19892427
- [Background] Sayed-Tabatabaei FA, Oostra BA, Isaacs A, van Duijn CM, Witteman JC. ACE polymorphisms. Circ Res. 2006 May 12;98(9):1123-33. doi: 10.1161/01.RES.0000223145.74217.e7. PMID 16690893
- [Background] Wuhl E, Witte K, Soergel M, Mehls O, Schaefer F; German Working Group on Pediatric Hypertension. Distribution of 24-h ambulatory blood pressure in children: normalized reference values and role of body dimensions. J Hypertens. 2002 Oct;20(10):1995-2007. doi: 10.1097/00004872-200210000-00019. PMID 12359978
- [Background] Soergel M, Kirschstein M, Busch C, Danne T, Gellermann J, Holl R, Krull F, Reichert H, Reusz GS, Rascher W. Oscillometric twenty-four-hour ambulatory blood pressure values in healthy children and adolescents: a multicenter trial including 1141 subjects. J Pediatr. 1997 Feb;130(2):178-84. doi: 10.1016/s0022-3476(97)70340-8. PMID 9042117
- [Background] ESCAPE Trial Group; Wuhl E, Trivelli A, Picca S, Litwin M, Peco-Antic A, Zurowska A, Testa S, Jankauskiene A, Emre S, Caldas-Afonso A, Anarat A, Niaudet P, Mir S, Bakkaloglu A, Enke B, Montini G, Wingen AM, Sallay P, Jeck N, Berg U, Caliskan S, Wygoda S, Hohbach-Hohenfellner K, Dusek J, Urasinski T, Arbeiter K, Neuhaus T, Gellermann J, Drozdz D, Fischbach M, Moller K, Wigger M, Peruzzi L, Mehls O, Schaefer F. Strict blood-pressure control and progression of renal failure in children. N Engl J Med. 2009 Oct 22;361(17):1639-50. doi: 10.1056/NEJMoa0902066. PMID 19846849
- [Background] Knoll GA, Cantarovitch M, Cole E, Gill J, Gourishankar S, Holland D, Kiberd B, Muirhead N, Prasad R, Tibbles LA, Treleaven D, Fergusson D. The Canadian ACE-inhibitor trial to improve renal outcomes and patient survival in kidney transplantation--study design. Nephrol Dial Transplant. 2008 Jan;23(1):354-8. doi: 10.1093/ndt/gfm574. Epub 2007 Sep 10. PMID 17848393
- [Background] Cooper WO, Hernandez-Diaz S, Arbogast PG, Dudley JA, Dyer S, Gideon PS, Hall K, Ray WA. Major congenital malformations after first-trimester exposure to ACE inhibitors. N Engl J Med. 2006 Jun 8;354(23):2443-51. doi: 10.1056/NEJMoa055202. PMID 16760444
- [Background] Urbina E, Alpert B, Flynn J, Hayman L, Harshfield GA, Jacobson M, Mahoney L, McCrindle B, Mietus-Snyder M, Steinberger J, Daniels S; American Heart Association Atherosclerosis, Hypertension, and Obesity in Youth Committee. Ambulatory blood pressure monitoring in children and adolescents: recommendations for standard assessment: a scientific statement from the American Heart Association Atherosclerosis, Hypertension, and Obesity in Youth Committee of the council on cardiovascular disease in the young and the council for high blood pressure research. Hypertension. 2008 Sep;52(3):433-51. doi: 10.1161/HYPERTENSIONAHA.108.190329. Epub 2008 Aug 4. No abstract available. PMID 18678786
- [Derived] Trachtman H, Frymoyer A, Lewandowski A, Greenbaum LA, Feig DI, Gipson DS, Warady BA, Goebel JW, Schwartz GJ, Lewis K, Anand R, Patel UD; Best Pharmaceuticals for Children Act-Pediatric Trials Network Administrative Core Committee. Pharmacokinetics, Pharmacodynamics, and Safety of Lisinopril in Pediatric Kidney Transplant Patients: Implications for Starting Dose Selection. Clin Pharmacol Ther. 2015 Jul;98(1):25-33. doi: 10.1002/cpt.127. Epub 2015 May 2. PMID 25807932
- See also: Pediatric Trials Network (PTN) — http://bpca.nichd.nih.gov/clinical/network/index.cfm
- See also: The Eunice Kennedy Shriver National Institute of Child Health and Human — http://www.nichd.nih.gov/
- See also: Information about Lisinopril — http://www.nlm.nih.gov/medlineplus/druginfo/meds/a692051.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low Dose: Lisinopril | Medium Dose: Lisinopril | High Dose: Lisinopril
Started | 13 | 10 | 3
Completed | 12 | 8 | 2
Not Completed | 1 | 2 | 1
Not completed — Insufficient PK sampling | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose: Lisinopril | Medium Dose: Lisinopril | High Dose: Lisinopril | Total
Number analyzed (Participants) | 12 | 8 | 2 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.9 (2.3) | 13.0 (3) | 9.5 (3.5) | 13.8 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 1 | 7
  Male | 8 | 6 | 1 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 4 | 0 | 7
  White | 7 | 2 | 2 | 11
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 12 | 8 | 2 | 22
Estimated glomerular filtration rate (eGFR) [Mean (Standard Deviation); unit: ml/min per 1.73m^2] — Estimated glomerular filtration rate (eGFR) calculated by modified Schwartz formula [=0.413 x Length (cm)/serum creatinine (mg/dl)].
  Note: text verified with protocol on 4/2/15 as '413xLength'. Added spaces for clarification.
  ml/min per 1.73m^2 | 72.5 (25.7) | 62 (16.7) | 89.3 (44.4) | 70.2 (24.4)
Time since transplant [Mean (Standard Deviation); unit: years] | 4.8 (4.7) | 4.9 (3.4) | 0.9 (0.4) | 4.5 (4.1)
Ethnicity [Number; unit: participants]
  Hispanic/Latino | 2 | 2 | 0 | 4
  Non-hispanic/non-latino | 10 | 6 | 2 | 18
Weight [Mean (Standard Deviation); unit: kg] | 56.8 (19.4) | 50.2 (28.7) | 23.1 (3.0) | 51.3 (23.8)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK) - Area Under the Plasma Concentration-time Curve (AUC)
Description: At the Day 14 (±3 days) visit, blood (1 mL) will be collected at 0 hour (pre-dose) and at 1, 2, 4, 5, 8, 12 and 24 hours post-lisinopril dose for determination of AUC. Geometric mean was calculated from all measurements.
Time Frame: Day 14 (+/- 3 days) of lisinopril therapy at hours 0 (pre-dose) and 1,2,4,5,8,12 and 24 hrs after dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Low Dose: Lisinopril | Medium Dose: Lisinopril | High Dose: Lisinopril
Number analyzed (Participants) | 12 | 8 | 2
ng*h/mL | 298 (46.5) | 640 (28.6) | 702 (66.4)

2. Primary Outcome: PK - Maximum Observed Concentration of Drug in Plasma (Cmax)
Description: At the Day 14 (±3 days) visit, blood (1 mL) will be collected at 0 hour (pre-dose) and at 1, 2, 4, 5, 8, 12 and 24 hours post-lisinopril dose for determination of Cmax. Geometric mean was calculated from all measurements.
Time Frame: Day14 (+/- 3 d) of dose at 0 hour and 1, 2, 4, 5, 8, 12, and 24 hrs after dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | Low Dose: Lisinopril | Medium Dose: Lisinopril | High Dose: Lisinopril
Number analyzed (Participants) | 12 | 8 | 2
ng/ml | 20.9 (41.2) | 47.7 (25.1) | 58.0 (41.2)

3. Secondary Outcome: Change in Potassium Level From Baseline in Lisinopril-naive Participants
Description: Potassium values will be obtained at Baseline and Day 14 prior to the final dose of study drug. Mean calculated from the two measurements.
Time Frame: At baseline visit and Day 14 prior to final study dose.
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Low Dose: Lisinopril | Medium Dose: Lisinopril | High Dose: Lisinopril
Number analyzed (Participants) | 6 | 6 | 3
mEq/L | 0.1 (0.3) | -0.3 (0.6) | 0.3 (0.5)

4. Secondary Outcome: Worse Post-dose Decrease in Estimated Glomerular Filtration Rate (eGFR) From Baseline in Lisinopril-naive Participants
Description: The eGFR at entry will need to be ≥ 30 ml/min/1.73m^2 to minimize concerns about an acute angiotensin-converting enzyme inhibitors (ACE-I)-mediated reduction in kidney function. eGFR ratio was computed from the worst post-dose value divided by the Baseline value.
Time Frame: Baseline to Day 14 (+/- 3 days)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Low Dose: Lisinopril | Medium Dose: Lisinopril | High Dose: Lisinopril
Number analyzed (Participants) | 6 | 6 | 3
ratio | 1 (14) | 1.02 (10) | 0.89 (14)

5. Primary Outcome: PK - Time of the Maximum Observed Concentration in Plasma (Tmax)
Description: At the Day 14 (±3 days) visit, blood (1 mL) will be collected at 0 hour (pre-dose) and at 1, 2, 4, 5, 8, 12 and 24 hours post-lisinopril dose for determination of plasma lisinopril concentration. Medium was calculated from all measurements.
Time Frame: Day 14 (+/- 3 d) of dose at 0 hour and 1, 2, 4, 5, 8, 12, and 24 hrs after dose
Measure: Median (Full Range); unit: hours
Arm/Group | Low Dose: Lisinopril | Medium Dose: Lisinopril | High Dose: Lisinopril
Number analyzed (Participants) | 12 | 8 | 2
hours | 5.0 [4.0 to 8.1] | 5.0 [4.0 to 8.0] | 4.5 [4.0 to 5.0]

6. Primary Outcome: PK - Oral Clearance (CL/F)
Description: At the Day 14 (±3 days) visit, blood (1 mL) will be collected at 0 hour (pre-dose) and at 1, 2, 4, 5, 8, 12 and 24 hours post-lisinopril dose for determination of CL/F. Geometric mean was calculated from all measurements.
Time Frame: Day 14 (+/- 3 d) of dose at 0 hour and at 1, 2, 4, 5, 8, 12, and 24 hrs after dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h/70 kg
Arm/Group | Low Dose: Lisinopril | Medium Dose: Lisinopril | High Dose: Lisinopril
Number analyzed (Participants) | 12 | 8 | 2
L/h/70 kg | 17.9 (61.2) | 18.6 (34.4) | 32.8 (54.1)

7. Primary Outcome: PK Renal Clearance (CLrenal)
Description: At the Day 14 (±3 days) visit, blood (1 mL) will be collected at 0 hour (pre-dose) and at 1, 2, 4, 5, 8, 12 and 24 hours post-lisinopril dose for determination of CLrenal. Geometric mean was calculated from all measurements.
Time Frame: Day 14 (+/- 3 d) of dose at 0 hour and 1, 2, 4, 5, 8, 12, and 24 hrs after dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h/70 kg
Arm/Group | Low Dose: Lisinopril | Medium Dose: Lisinopril | High Dose: Lisinopril
Number analyzed (Participants) | 12 | 8 | 2
L/h/70 kg | 3.4 (60.4) | 3.4 (46.0) | 6.8 (94.4)

8. Primary Outcome: Number of Adverse Events (AEs) and Serious Adverse Events (SAEs) During/After Study Drug Administration
Description: Number of Adverse Events (AEs) related and not related to study drug; number of Serious Adverse Events (SAEs) related and not related to study drug
Time Frame: First dose of study drug to 30 days after final study visit for AEs and until resolution for SAEs
Measure: Number; unit: events
Groups:
- Lisinopril-naive: These protocol participants were not randomized. Instead, the older age group (7-17 years) were first enrolled consecutively into each dose level, starting with the lowest dose level (0.1 mg/kg per day). After enrollment is complete in the low dose level for an eGFR strata, enrollment will commence for the intermediate (0.2 mg/kg per day) dosage in that strata, followed by the high (0.4 mg/kg per day) dosage level. Enrollment for the 2-6 years age group did not begin until enrollment in the older age group (7-17 years) for the low and intermediate dosage level at each eGFR strata is complete.
- Lisinopril Standard of Care (SOC): These protocol participants were enrolled and continued on the lisinopril dose prescribed as standard of care. They were assigned to the appropriate eGFR and dose level stratum (rounding to the closest dose level). Since the lisinopril dose was assigned based on standard of care, a patient was enrolled without regard to open/closed status of the dose stratum in this group. Therefore, over enrollment of a specific dose and eGFR stratum was allowed for participants enrolled he the Lisinopril-naive group to accommodate these valuable low-risk participants already taking lisinopril.
Arm/Group | Lisinopril-naive | Lisinopril Standard of Care (SOC)
Number analyzed (Participants) | 15 | 11
events
  AEs | 12 | 12
  AE related to study drug | 5 | 0
  AEs not related to study drug | 7 | 12
  SAE | 1 | 0
  SAE not related to study drug | 1 | 0

9. Secondary Outcome: Largest eGFR Percent Decrease From Baseline in Lisinopril-naive Participants
Description: The eGFR at entry will need to be ≥ 30 ml/min/1.73m^2 to minimize concerns about an acute angiotensin-converting enzyme inhibitor (ACEI) mediated reduction in kidney function.
  Largest eGFR percent decrease from baseline reported in results section.
Time Frame: Baseline to Day 14 (+/- 3 days)
Measure: Number; unit: percentage
Arm/Group | Low Dose: Lisinopril | Medium Dose: Lisinopril | High Dose: Lisinopril
Number analyzed (Participants) | 6 | 6 | 3
percentage | 15 | 12 | 21

10. Secondary Outcome: Change in Urine Protein/Creatinine From Baseline in Lisinopril-naive Participants.
Description: Change in urine protein/creatinine obtained as follows: Mean change (worst post-dose from baseline) presented for urine protein/creatinine ratio. Geometric mean of the ratio (worst post-dose / baseline with Geometric Coefficient of Variation percent (CV%) and greatest decrease presented for eGFR by dose group. Two patients in the high dose group had an evaluable urine protein/creatinine change.
Time Frame: Baseline to worst post-dose before Day 14 (+/- 3 days)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/mg
Arm/Group | Low Dose: Lisinopril | Medium Dose: Lisinopril | High Dose: Lisinopril
Number analyzed (Participants) | 6 | 6 | 3
mg/mg | -0.45 (0.6) | -0.08 (0.15) | -0.74 (1.37)

11. Secondary Outcome: Change in Diastolic Blood Pressure From Baseline in Lisinopril-naive Participants
Description: Ambulatory blood pressure readings were measured during the baseline/pre-study dose period using a SpaceLabs (Redmond, WA) device at home to avoid the confounding effects of venipuncture and abnormal sleep pattern.
  Another blood pressure reading was performed at 1 day before the final dose of lisinopril (day before the last scheduled visit).
  The mean of these measurements was calculated.
Time Frame: Baseline to Day 14 (+/-3 days)
Population: Change in diastolic blood pressure from baseline is reported here for lisinopril-naive participants (not the standard of care group which are reported separately).
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Low Dose: Lisinopril | Medium Dose: Lisinopril | High Dose: Lisinopril
Number analyzed (Participants) | 6 | 6 | 3
mmHg
  eGFR 30-59 ml/min per 1.73m^2 (n=3, 1, 0) | -4.0 (20) | 7.0 (0) | NA (NA) — no participants in this category
  eGFR >=60 ml/min per 1.73m^2 (n=3, 5, 3) | -9.0 (7.5) | -6.0 (6.7) | -4.0 (5.3)

12. Secondary Outcome: Change in Systolic Blood Pressure From Baseline in Lisinopril-naive Participants
Description: Ambulatory blood pressure readings were measured during the baseline/pre-study dose period using a SpaceLabs (Redmond, WA) device at home to avoid the confounding effects of venipuncture and abnormal sleep pattern.
  Another blood pressure reading was performed at 1 day before the final dose of lisinopril (day before the last scheduled visit).
  The mean from these measurements was calculated.
Time Frame: Baseline to Day 14 (+/- 3 days)
Population: Change in systolic blood pressure from baseline is reported here for lisinopril-naive participants (not the standard of care (SOC) group which are reported separately).
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Low Dose: Lisinopril | Medium Dose: Lisinopril | High Dose: Lisinopril
Number analyzed (Participants) | 6 | 6 | 3
mmHg
  eGFR 30-59 ml/min per 1.73m2 (n=3, 1, 0) | -5.0 (11.4) | -6.0 (0) | NA (NA) — no participants in this category
  eGFR >+60 ml/min per 1.732 (n=3, 5, 3) | -6.7 (4.0) | -8.8 (11.7) | -11.3 (2.1)

13. Secondary Outcome: Change in Systolic Blood Pressure (BP) From Baseline in Lisinopril SOC Group
Description: Lisinopril SOC participants were not given the ambulatory blood pressure machine to obtain readings at home, as was the Lisinopril-naive participants. Instead BP measurements were obtained during screening visit and compared to the Day 14 to 40 visit measurements. Note: these participants were not required to attend a Day 14 (+/-3 day visit) but did need to attend sometime between Day 14 to Day 40 (inclusive). The mean of these blood pressure measurements was calculated.
Time Frame: Screening to Day 14 to 40
Population: Change in systolic blood pressure from baseline is reported here for lisinopril SOCparticipants (not the Lisinopril-naive group which are reported separately).
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Low Dose: Lisinopril | Medium Dose: Lisinopril | High Dose: Lisinopril
Number analyzed (Participants) | 7 | 4 | 0
mmHg
  eGFR 30-59 ml/min per 1.73m2 (n=2, 2, 0) | -6.0 (17) | -1.0 (4.2) |
  eGFR >=60 ml/min per 1.73m2 (n=5, 2, 0) | 6.4 (6.9) | -1.0 (0) |

14. Secondary Outcome: Change in Diastolic Blood Pressure From Baseline in Lisinopril SOC Group
Description: Lisinopril SOC participants were not given the ambulatory blood pressure machine to obtain readings at home, as was the Lisinopril-naive participants. Instead BP measurements were obtained during screening visit and compared to the Day 14 to 40 visit measurements (note: the participants were not required to attend a Day 14 (+/-3 day visit) but did need to attend sometime between Day 14 to Day 40. The mean from the blood pressure measurements was calculated.
Time Frame: Screening to Day 14 to 40
Population: Change in diastolic blood pressure from baseline is reported here for lisinopril SOCparticipants (not the Lisinopril-naive group which are reported separately).
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Low Dose: Lisinopril | Medium Dose: Lisinopril | High Dose: Lisinopril
Number analyzed (Participants) | 7 | 4 | 0
mmHg
  eGFR 30-59 ml/min per 1.73m2 (n=2, 2, 0) | -6.0 (5.7) | -6.5 (9.2) |
  eGFR >=60 ml/min per 1.73m2 (n=5, 2, 0) | 3.4 (14.0) | -3.0 (0) |

ADVERSE EVENTS:
Arm/Group | Low Dose: Lisinopril | Medium Dose: Lisinopril | High Dose: Lisinopril
Serious Adverse Events (participants affected / at risk) | 0/12 | 1/8 | 0/2
Other Adverse Events (participants affected / at risk) | 5/12 | 4/8 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose: Lisinopril (N=12) | Medium Dose: Lisinopril (N=8) | High Dose: Lisinopril (N=2)
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose: Lisinopril (N=12) | Medium Dose: Lisinopril (N=8) | High Dose: Lisinopril (N=2)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0
Retching (Gastrointestinal disorders) | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Infusion site extravasation (General disorders) | 1 | 0 | 0
Infusion site pain (General disorders) | 1 | 0 | 0
Infusion site pruritus (General disorders) | 1 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 1
Hemoglobin decreased (Investigations) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 2 | 0
Headache (Nervous system disorders) | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No